CLINICAL TRIAL: NCT06641180
Title: A Phase 3, Randomized, Modified Double-blind, 2-arm Study to Evaluate the Immunogenicity and Safety of High-Dose Inactivated Influenza Vaccine (IIV-HD) Compared With a Standard-dose Inactivated Influenza Vaccine (IIV-SD) in Participants 50 Through 64 Years of Age.
Brief Title: Study to Evaluate Immunogenicity and Safety of a High-Dose Influenza Vaccine in Adults 50 Through 64 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QHD00042; U1111-1305-7370 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind:
  * Participants, Sponsor study staff*, investigators, and study site staff will not know which study vaccine is administered during the study conduct
  * Dedicated study site staff who prepare/administer the study interventions and are not involved in the safety evaluation will know which study vaccine is administered.
    * Select sponsor staff will be unblinded after the code break for primary completion analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IIV-HD (Experimental): Participants will receive a single intramuscular (IM) injection of IIV-HD at Day 1
  Interventions: Biological: High-Dose trivalent influenza vaccine (Split virion, Inactivated)
- IIV-SD (Active Comparator): Participants will receive a single intramuscular (IM) injection of IIV-SD at Day 1
  Interventions: Biological: Standard-dose trivalent influenza vaccine (Split virion, Inactivated)

INTERVENTIONS:
Biological: High-Dose trivalent influenza vaccine (Split virion, Inactivated) — Liquid suspension for intramuscular injection
  Arms: IIV-HD
Biological: Standard-dose trivalent influenza vaccine (Split virion, Inactivated) — Liquid suspension for intramuscular injection
  Arms: IIV-SD

SUMMARY:
The purpose of this study is to evaluate Immunogenicity and Safety of a High-Dose (HD) Influenza Vaccine (IV) in Adults 50 through 64 Years of Age.

DETAILED DESCRIPTION:
The study duration will be approximately 180 days (+ 14 days).

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 to 64 years on the day of inclusion.
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, or surgically sterile.

OR

* Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 4 weeks after study intervention administration.
* A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) at enrollment before the first dose of study intervention.

  * Informed consent form has been signed and dated.
  * Able to attend all scheduled visits and to comply with all study procedures.

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Personal or family history of Guillain-Barré Syndrome (GBS).
* Known systemic hypersensitivity to any of the study intervention components (Section 1.1, Section 6.1), or history of a life-threatening reaction to the study intervention used in the study or to a product containing any of the same substances.
* Self-reported thrombocytopenia, contraindicating intramuscular injection, based on investigator's judgment.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular injection, based on investigator's judgment.
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of study intervention administration. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion.
* Receipt of any vaccine in the 4 weeks preceding the study intervention administration or planned receipt of any vaccine prior to the second blood drawing (ie. approximately 4 weeks after the study intervention administration).
* Previous vaccination against influenza in the previous 6 months with an investigational or marketed vaccine.
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months.
* Participation at the time of study enrollment (or in the 4 weeks preceding the first study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Deprived of freedom by an administrative or court order, or being in an emergency setting, or hospitalized involuntarily.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie.

parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1180 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Geometric mean titers (GMTs) against influenza vaccine antibodies (Ab) | Day 1 and Day 29
  GMTs of anti-influenza antibodies were measured using hemagglutination inhibition (HAI) assay for 3 influenza virus strains: A/H1N1, A/H3N2, and B/Victoria lineage.
Percentage of participants with seroconversion for influenza vaccine antibodies | Day 29
  Anti-influenza antibodies will be measured using HAI assay for 3 influenza virus strains: A/H1N1, A/H3N2, and B/Victoria lineage. Seroconversion status 28 days after vaccination (ie, preinjection Ab titer < 10 [1/dil] at Day 1 and post-injection Ab titer≥ 40 [1/dil] at Day 29 or preinjection Ab titer ≥ 10 [1/dil] at Day 1 and a ≥ 4-fold increase in titer [1/dil] at Day 29).

SECONDARY OUTCOMES:
Geometric Mean of Individual Titer Ratio (GMTR) | Day 1 and Day 29
  GMTRs will be measured using HAI assay for 3 influenza virus strains: A/H1N1, A/H3N2, and B/Victoria lineage. Individual HAI antibody titer ratio Day 29/Day 1.
Percentage of participants with detectable HAI titer (HAI titer ≥ 10 [1/dil]) | Day 1 and Day 29
  Anti-influenza antibodies will be measured using HAI assay for 3 influenza virus strains: A/H1N1, A/H3N2, and B/Victoria lineage. Percentage of participants with HAI antibody titer >=10 (1/dil)
Percentage of participants with HAI titer ≥ 40 (1/dil) | Day 29
  Anti-influenza antibodies will be measured using HAI assay for 3 influenza virus strains: A/H1N1, A/H3N2, and B/Victoria lineage. Percentage of participants with HAI antibody titers ≥ 40 (1/dil)
Number of participants with immediate adverse events (AEs) | Within 30 minutes after vaccination
  Immediate events are recorded to capture medically relevant unsolicited systemic AEs which occur within the first 30 minutes after vaccination.
Number of participants with solicited injection site reactions | Up to 7 days after vaccination
  Solicited injection site reactions (pre-listed in the participant diary and CRF)
Number of participants with solicited systemic reaction | Up to 7 days after vaccination
  Solicited systemic reactions (pre-listed in the participant diary and CRF)
Number of participants with unsolicited AEs | Up to 28 days after vaccination
  An unsolicited AE is an observed AE that does not fulfill the conditions of solicited reactions, ie, pre-listed in the CRF in terms of diagnosis and onset window post-vaccination.
Number of participants with medically attended adverse events (MAAEs) | Throughout the study, approximately 180 days
  An MAAE is a new-onset or a worsening of a condition that prompts the participant or participant's parent(s)/legally acceptable representative(s) to seek unplanned medical advice at a physician's office or Emergency Department.
Number of participants with adverse events of special interest (AESIs) | Throughout the study, approximately 180 days
  An adverse event of special interest (serious or non-serious) is one of scientific and medical concern specific to the Sponsor's study intervention or program, for which ongoing monitoring and rapid communication by the investigator to the Sponsor can be appropriate.
Number of participants with serious adverse events (SAEs) | Throughout the study, approximately 180 days
  A SAE is defined as any adverse event that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was other medically important event.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - CenExel CNS- Site Number : 8400005, Los Alamitos, California
  - Alliance for Multispeciality Research - Fort Myers- Site Number : 8400019, Fort Myers, Florida
  - Research Centers of America - Hollywood- Site Number : 8400010, Hollywood, Florida
  - IACT Health - Columbus - Talbotton Road- Site Number : 8400011, Columbus, Georgia
  - Cenexel IRA - iResearch Atlanta- Site Number : 8400007, Decatur, Georgia
  - The Hope Clinic of Emory Vaccine Center- Site Number : 8400017, Decatur, Georgia
  - Centricity Research - Rincon- Site Number : 8400012, Rincon, Georgia
  - Cenexel IRS - iResearch Savannah- Site Number : 8400008, Savannah, Georgia
  - Alliance for Multispeciality Research - Newton- Site Number : 8400003, Newton, Kansas
  - Alliance for Multispeciality Research - Lexington- Site Number : 8400002, Lexington, Kentucky
  - CBH Health - Gaithersburg- Site Number : 8400004, Gaithersburg, Maryland
  - Hassman Research Institute - Berlin- Site Number : 8400006, Berlin, New Jersey
  - Centricity Morehead- Site Number : 8400014, Morehead City, North Carolina
  - Centricity New Bern- Site Number : 8400015, New Bern, North Carolina
  - Aventiv Research Columbus- Site Number : 8400016, Columbus, Ohio
  - Kaiser Permanente Center for Health Research- Site Number : 8400018, Portland, Oregon
  - Alliance for Multispecialty Research - Volunteer Research Group- Site Number : 8400001, Knoxville, Tennessee
  - JBR Clinical Research- Site Number : 8400009, Salt Lake City, Utah
  - Centricity Research - Suffolk Primary Care - Centricity - PPDS- Site Number : 8400013, Suffolk, Virginia
  - Kaiser Permanente Washington- Site Number : 8400024, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: QHD00042 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26147&tenant=MT_SNY_9011